CLINICAL TRIAL: NCT03075995
Title: To Discuss the Best Mode for Taking Lapatinib Under the Influence of the Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xu fei, Associate Senior Doctor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU002
Record Dates: First submitted 2017-03-02; First posted 2017-03-09 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: lapatinib; steady state plasma concentration; high-fat breakfast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: It's divided into two stages.For the first stage,the subjects take lapatinib on an empty stomach,the steady state plasa concentration is examined on the 9th and 10th days after lapatinib is administered.The second stage,the subject take lapatinib with hight-fat breakfast,the steady state plasa concentration is examined as the first stage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lapatinib administered with hight-fat breakfast (Experimental)
  Interventions: Other: hight-fat breakfast

INTERVENTIONS:
Other: hight-fat breakfast — It's divided into two stages.For the first stage,the subjects take lapatinib on an empty stomach,the steady state plasa concentration is examined on the 9th and 10th days after lapatinib is administered.The second stage,the subject take lapatinib with hight-fat breakfast,the steady state plasa concentration is examined as the first stage.

SUMMARY:
Food can make a big difference on the bioavailability of lapatinib in breast cancer patients,and fatty food can increase the lapatinib bioavailability.By examine the steady blood drug concentration in the same individual at different treatment mode for lapatinib,emptiness or taken with fatty food,discuss the best mode of taking lapatinib with fatty food.

DETAILED DESCRIPTION:
Metastatic breast cancer is the leading cause of cancer-related death among women worldwide ,those overexpress the HER2 are associated with a higher risk. Lapatinib is approved for use to treat advanced metastatic breast cancer. The pharmacokinetic parameters of lapatinib have been characterized previously.It can reach steady state concentration after 6 or 7 days oral dosing, but the bioavailability is very different between different patients. The effect of food on lapatinib pharmacokinetics in humans was first examined in 19 healthy participants who were given single 100-mg doses with a high-fat breakfast. Food caused a 60% increase in the relative bioavailability of lapatinib.Another test showed that the bioavailability of lapatinib was 3 times more in low-fat diet than in emptiness.

Some investigators think that it can change the mode for taking lapatinib with food or without food to enhance the absorption.It may decrease the oral dose but the lapatinib can reach the same steady state concentration,so it can achieve maximum economic benefits.

By continuous change for lapatinib and fat diet, The change of lapatinib pharmacokinetic is lack of discussion. If the adverse reactions increase since the absorption of lapatinib increase, the existing research data are still lacking.

The trial By examine the steady blood drug concentration in the same individual at different treatment mode for lapatinib, emptiness or taken with fatty food, discuss the best mode of taking lapatinib with fatty food.

ELIGIBILITY:
Inclusion Criteria:

1. Advance breast cancer with her2 positive
2. The patients are ready to use or using lapatinib for tumor treatment, and plans to keep the treatment for at least a month
3. The ECOG score is 0 to 2
4. hemoglobin≥ 9 gm/dL
5. serum albumin concentration is normal
6. ALT / AST / bilirubin<1.5UL
7. creatinine clearance rate≥ 40 mL/min
8. signed ICF

Exclusion Criteria:

1. Pregnancy or Pregnancy
2. Stomach absorption dysfunction
3. Difficulty in taking fatty food
4. Severe heart disease or medical condition

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
the Best Mode for Takeing Lapatinib | 20 days
  by examined the steady state plasa concentration of Lapatinib ,determine which is the best way to take lapatinib,with high-fat breakfast or on an empty stomach

CONTACTS AND LOCATIONS:
Overall Officials: Fei Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No